CLINICAL TRIAL: NCT04841252
Title: Classification of Breast Masses Based on Visco-elastic Properties Using SAVE Method
Acronym: SAVE
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Azra Alizad, Principal Investigator, Mayo Clinic
Other Study IDs: 12-009399
Record Dates: First submitted 2021-04-06; First posted 2021-04-12 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: FDA approved GE LOGIQ E9 (LE9) ultrasound — Ultrasound
Device: Alpinion clinical ultrasound machine — Ultrasound

SUMMARY:
The purpose of this research is to conduct a clinical study to evaluate the efficacy of a noninvasive and quantitative tool for classification/diagnosis of breast masses. The main objective of this proposal is to test the SAVE (Sub-Hertz Analysis of Visco-Elasticity) method on a patient population of sufficient size to determine the sensitivity and specificity for malignant-benign discrimination of breast masses.

DETAILED DESCRIPTION:
Subject will sit or lie back on an examination bed. The investigators will use an ultrasound scanner to collect sonographic imaging data from the breast. For this purpose the investigators may use a clinical scanner such as Supersonics Aixplorer or similar or a research ultrasound machine such as Verasonics (this machine has been use in other Mayo IRB approved protocols such as IRB 11-001953). The ultrasound probe will be placed on the breast to visualize the mass. The probe will be pressed with a constant force for a period of 10-40 seconds. During this time ultrasound data will be recorded by the ultrasound scanner.

To keep the probe pressed on the breast with a constant force, the user may hold the probe by hand and press it steadily against the breast at constant force. This force is only a few Newtons (approximately half a Kg weight) which should be quite tolerable for a typical patient. Alternatively, the investigators may use an automated "actuator" to hold the probe steady and press it against the breast at a constant force to the same level. The reason for pressing the breast is to determine how the breast tissue gradually deforms; therefore this method to some extent simulates breast palpation.

The time needed to scan a subject for this study is short (a few minutes to set up, and about 10-40 seconds to scan). It will take approximately 20 minutes to complete the study. The scan can be done at the time of clinical breast sonography. The subject may be asked to hold her breath during the scan time if possible.

The investigators call this method "Sub-Hertz Analysis of Visco-Elasticity (SAVE)".

To facilitate subject access and shorten patient participation time, the investigator may station our system in the Breast Imaging area where routine clinical imaging procedures are performed.

The investigators may also use the FDA approved GE LOGIQ E9 (LE9) ultrasound system to quantify and image the stiffness of the breast lesion and compare the results to those obtained by the investigational device.

The investigators may also use the Alpinion clinical ultrasound machine, both FDA approved clinical format ECUBE 12 and non FDA approved ECUBE 12R format to acquire ultrasound images.

ELIGIBILITY:
Inclusion Criteria:

* Females in age range between 18 and up who have a breast lesion that may or may not be suspicious for breast cancer, and are referred for Radiological investigation.

Exclusion Criteria:

* No history of mastectomy or implants, or having any condition that does not allow proper use of our imaging devices.
* Only include patients with masses detectable under ultrasound.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Females in age range between 18 and up who have a breast lesion that may or may not be suspicious for breast cancer, and are referred for Radiological investigation.
Study Population: Females in age range between 18 and up who have a breast lesion that may or may not be suspicious for breast cancer
Sampling Method: Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2012-12-19 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

PRIMARY OUTCOMES:
Determine the efficacy of the SAVE method by correlating its results with pathology in a pathology in a population of patients with suspicious breast masses. | Before biopsy or at least 2 weeks post biopsy
  Assessed using a two-phase design. The first phase will be the development aspects to determine a candidate threshold for T1 that produces Optimal diagnostic accuracy as quantified by the largest diagnostic odds ratio.
  The second phase of the study will be to apply this candidate threshold to the validation sample enrolled as a part of the specific aim to ensure diagnostic utility. For both phases of the analysis, overall diagnostic accuracy will be quantified by the area under the receiver operating characteristics (ROC) curve.
Determine the efficacy of SAVE method in classifying non-specific masses in a group of breast patients on the follow-up list. | Before biopsy or at least 2 weeks post biopsy
  The threshold determined in Aim 1 will be applied to the patients in this sample to calculate the diagnostic performance

CONTACTS AND LOCATIONS:
Overall Officials: Azra Alizad, M.D., Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials